CLINICAL TRIAL: NCT06476561
Title: The Impact of Sociodemographic, Psychological, and Quality of Life Factors on Dual-Task Performance in Elderly Individuals: A Cross-Sectional Study in Iraq
Brief Title: Impact of Sociodemographic, Psychological, and Quality of Life Factors on Dual-Task Performance in Elderly Iraqis
Acronym: SociQ-DT
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Assoc. Prof., Çankırı Karatekin University
Other Study IDs: 1bd259b9391040ed].
Record Dates: First submitted 2024-06-19; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Cognitive Dysfunction; Motor Skills Disorders; Aging
Keywords: Dual-Task Performance; Elderly; Cognitive Function; Motor Skills; Quality of Life; Physical Health
MeSH Terms: conditions — Cognitive Dysfunction; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Participants in Iraq: This study group consists of community-dwelling elderly individuals aged 60 and above residing in Najaf, Iraq. The participants are healthy and do not have severe physical or mental health conditions. They are evaluated to understand how sociodemographic, psychological, and quality of life factors influence their dual-task performance, which includes both cognitive and motor functions. The study aims to provide insights into factors affecting their ability to perform dual tasks, contributing to the development of targeted interventions and policies for improving the quality of life and care for Iraq's aging population.
  Interventions: Other: - Sociodemographic Assessment - Psychological Assessment - Quality of Life Assessment - D

INTERVENTIONS:
Other: - Sociodemographic Assessment - Psychological Assessment - Quality of Life Assessment - D — The study involves several assessments to evaluate the impact of various factors on dual-task performance in elderly individuals:
  1. Sociodemographic Assessment: Collection of data on age, gender, education, income, marital status, and other relevant factors.
  2. Psychological Assessment: Use of the Depression Anxiety Stress Scales-21 (DASS-21) to measure levels of depression, anxiety, and stress.
  3. Quality of Life Assessment: Utilization of the World Health Organization Quality of Life Brief Form (WHOQOL-BREF) to assess physical health, psychological health, social relationships, and environment.
  4. Dual-Task Performance Evaluation: Measurement of the ability to perform a cognitive task (counting backward by threes) simultaneously with a motor task (Nine-Hole Peg Test). The dual-task cost (DTC) is calculated to quantify the impact of cognitive load on motor performance.

SUMMARY:
This study investigates the impact of sociodemographic, psychological, and quality of life factors on dual-task performance in elderly individuals living in Iraq. Dual-task performance, the ability to perform two tasks simultaneously, is a crucial indicator of cognitive and motor functions in older adults. This research aims to understand how factors such as age, gender, education, income, mental health (depression, anxiety, and stress), mindfulness, and overall quality of life influence the ability of elderly individuals to manage dual tasks, which is essential for maintaining independence and preventing falls.

The study hypothesizes that better physical health and quality of life will be associated with improved dual-task performance, while higher levels of psychological distress may negatively impact this ability. Data were collected from 384 healthy community-dwelling elderly participants aged 60 and above in Najaf, Iraq, using validated tools such as the Depression Anxiety Stress Scales-21 (DASS-21), the Mindful Attention Awareness Scale (MAAS), and the World Health Organization Quality of Life Brief Form (WHOQOL-BREF). Dual-task performance was assessed through the Nine-Hole Peg Test (NHPT) combined with a cognitive task of counting backward by threes.

The findings from this study will provide valuable insights into the factors that affect cognitive and motor functions in the elderly, helping to inform the development of targeted interventions and policies aimed at improving the quality of life and care for Iraq's aging population. Understanding these influences is crucial for enhancing elderly care, preventing falls, supporting cognitive health, and informing policies to improve the quality of life for Iraq's aging population.

DETAILED DESCRIPTION:
This cross-sectional study aims to explore the impact of sociodemographic, psychological, and quality of life factors on dual-task performance in elderly individuals living in Najaf, Iraq. Dual-task performance is critical for assessing cognitive and motor functions, and understanding these influences is essential for enhancing elderly care, preventing falls, supporting cognitive health, and informing policies to improve the quality of life for Iraq's aging population.

Study Hypothesis:

The study hypothesizes that better physical health and quality of life will be associated with improved dual-task performance, while higher levels of psychological distress (depression, anxiety, and stress) will negatively impact this ability.

Participants:

The study includes 384 healthy community-dwelling participants aged 60 and above, recruited from various community centers, healthcare facilities, and local organizations in Najaf, Iraq. Inclusion criteria cover individuals irrespective of gender, marital status, education level, income, socioeconomic status, urban or rural residence, and employment status. Exclusion criteria include severe physical or mental health conditions, language barriers, severe communication issues, and unwillingness to participate. Cognitive status below the Mild Cognitive Impairment (MCI) limit based on evaluator observations also led to exclusion.

Data Collection Tools:

1. Depression Anxiety Stress Scales-21 (DASS-21): A 21-item scale assessing depression, anxiety, and stress, rated on a 4-point Likert scale.
2. Mindful Attention Awareness Scale (MAAS): A 15-item instrument measuring mindfulness, rated on a 6-point Likert scale.
3. World Health Organization Quality of Life - BREF (WHOQOL-BREF): A 26-item questionnaire measuring physical health, psychological health, social relationships, and environment.

Dual-Task Performance Assessment:

Participants' dual-task performance was evaluated using the Nine-Hole Peg Test (NHPT), where they place and remove nine pegs in a series of holes as quickly as possible. This motor task was combined with a cognitive task of counting backward by threes. Performance was assessed by comparing the time taken to complete the NHPT alone with the time taken while also performing the cognitive task.

Statistical Analysis:

Data were analyzed using SPSS version 23.0. Descriptive statistics summarized demographic characteristics and scale scores. Correlation analyses examined relationships between variables affecting dual-task performance. Pearson correlation coefficients were calculated for these analyses. Multivariate regression analyses were employed to isolate the independent effects of the variables on dual-task performance, with independent variables including demographic factors (age), DASS-21, MAAS, and WHOQOL-BREF scores. The regression model's goodness-of-fit was assessed using R-squared, adjusted R-squared, and F-statistic values. Regression coefficients, standard errors, and t-statistics tested the significance of predictors, with a significance level of \( p < 0.05 \) for all hypothesis tests. Data normality was evaluated using Kolmogorov-Smirnov and Shapiro-Wilk tests, confirming normal distribution. Missing data analysis ensured data integrity and completeness.

Sample Size Assessment:

A sample size of 384 participants was calculated to ensure a representative sample of the elderly population in Najaf, Iraq, with a 95% confidence level and a 5% margin of error.

Plan for Missing Data:

Missing data were addressed by determining if data were missing at random. Appropriate statistical methods were applied to handle missing data, ensuring the integrity of the dataset used in analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and above
* Healthy community-dwelling individuals
* Ability to understand and comply with study procedures
* Willingness to provide informed consent
* Residing in Najaf, Iraq

Exclusion Criteria:

* Severe physical health conditions
* Severe mental health conditions (e.g., severe depression, severe anxiety, schizophrenia)
* Cognitive status below the Mild Cognitive Impairment (MCI) limit
* Language barriers preventing understanding of study procedures
* Severe communication issues
* Unwillingness to participate
* Presence of consciousness disorders such as dementia
* Any condition that, in the opinion of the investigators, would interfere with the ability to complete the study or pose a risk to the participant's health

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: **Study Population Description:**
  The study population consists of healthy, community-dwelling elderly individuals aged 60 and above residing in Najaf, Iraq. Participants are recruited from various community centers, healthcare facilities, and local organizations within the city. The population includes individuals from diverse sociodemographic backgrounds, ensuring a representative sample of the elderly community in Najaf. The focus is on those who are generally healthy and capable of understanding and participating in the study procedures, excluding individuals with severe physical or mental health conditions or significant cognitive impairments.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Dual-Task Performance | The measurement is assessed at a single point in time during the participant's enrollment visit, immediately following the completion of both single-task and dual-task conditions.
  The primary outcome measure is the dual-task performance, assessed by the time taken to complete the Nine-Hole Peg Test (NHPT) while simultaneously performing a cognitive task of counting backward by threes.
  This metric characterizes the impact of cognitive load on motor performance, with higher DTC values indicating greater difficulty in managing dual tasks.

SECONDARY OUTCOMES:
Psychological Distress Levels | The measurement is assessed at a single point in time during the participant's enrollment visit, immediately following the completion of the DASS-21 questionnaire.
  Measurement of participants' levels of depression, anxiety, and stress using the Depression Anxiety Stress Scales-21 (DASS-21). Scores are calculated for each subscale (depression, anxiety, and stress) based on participants' responses, providing insight into the psychological well-being of the elderly population and its potential association with dual-task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyhun Türkmen, PhD, Principal Investigator — Çankırı Karatekin University Faculty of Health Sciences Department of Occupational Therapy
Locations (1):
- Ceyhun Türkmen, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) that underlie the results in the publication will be shared, including data dictionaries. This will ensure that other researchers can verify the findings and conduct further analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and additional supporting information will become available starting 6 months after the publication of the study results and will be accessible for a period of 5 years thereafter.
Access Criteria: IPD and supporting information will be shared with researchers who provide a methodologically sound proposal. Proposals should be directed to the principal investigator, Dr. Ceyhun Türkmen, and will be reviewed by the study's ethics committee. Data access will be granted for the purpose of replicating results or conducting further research on the same or related topics. Researchers will be required to sign a data use agreement before accessing the data.

REFERENCES:
- [Result] Abo M, Hamaguchi T. Effectiveness of a Dual-Task Intervention Involving Exercise and Vocalized Cognitive Tasks. J Clin Med. 2024 May 17;13(10):2962. doi: 10.3390/jcm13102962. PMID 38792503
- [Result] Mahmood KA, Saleh AM. Barriers and facilitators influencing access to and utilization of primary healthcare services in Kurdistan-region, Iraq: a cross-sectional study. Ann Med Surg (Lond). 2023 Jun 10;85(7):3409-3417. doi: 10.1097/MS9.0000000000000957. eCollection 2023 Jul. PMID 37427184
- [Result] Ali AM, Ahmed A, Sharaf A, Kawakami N, Abdeldayem SM, Green J. The Arabic Version of The Depression Anxiety Stress Scale-21: Cumulative scaling and discriminant-validation testing. Asian J Psychiatr. 2017 Dec;30:56-58. doi: 10.1016/j.ajp.2017.07.018. Epub 2017 Jul 18. PMID 28755630
- [Result] Baek JE, Hyeon SJ, Kim M, Cho HY, Hahm SC. Effects of dual-task resistance exercise on cognition, mood, depression, functional fitness, and activities of daily living in older adults with cognitive impairment: a single-blinded, randomized controlled trial. BMC Geriatr. 2024 Apr 24;24(1):369. doi: 10.1186/s12877-024-04942-1. PMID 38658827
- [Result] Bherer L, Erickson KI, Liu-Ambrose T. A review of the effects of physical activity and exercise on cognitive and brain functions in older adults. J Aging Res. 2013;2013:657508. doi: 10.1155/2013/657508. Epub 2013 Sep 11. PMID 24102028
- [Result] Bowen A, Wenman R, Mickelborough J, Foster J, Hill E, Tallis R. Dual-task effects of talking while walking on velocity and balance following a stroke. Age Ageing. 2001 Jul;30(4):319-23. doi: 10.1093/ageing/30.4.319. PMID 11509310